CLINICAL TRIAL: NCT06099639
Title: Medical Access Program for Patritumab Deruxtecan (HER3 DXd, U3-1402)
Brief Title: Medical Access Program for Patritumab Deruxtecan
Status: No longer available | Type: Expanded Access
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: U31402-0001-EAP-MA
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Epidermal Growth Factor Receptor (EGFR)-Mutated Non Small Cell Lung Cancer
Keywords: EGFR-mutated non small cell lung cancer; HER3 DXd; U3-1402
MeSH Terms: interventions — patritumab deruxtecan

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: HER3-DXd — 5.6 mg/kg Q3W [on Day 1 of each 21-day cycle]) infused IV over approximately 90 minutes
  Other Names: U3-1402

SUMMARY:
The purpose of this Medical Access Program is to provide access to HER3-DXd for eligible patients with NSCLC who, in their treating physician's opinion, have an unmet clinical need which cannot be treated with approved and commercially available drugs and who cannot enter a clinical trial prior to commercial availability.

DETAILED DESCRIPTION:
This is a Medical Access Program which will be available to adult patients in the US with metastatic or locally advanced EGFRm NSCLC who have received at least 2 prior systemic therapies, who have no alternative commercially available treatment options, and are not able to enter a clinical trial.

In this Medical Access Program, eligible patients will be treated with HER3-DXd and will continue to receive treatment until any of the following occurs:

* Disease progression
* Unacceptable toxicity
* The benefit-risk no longer favors the individual
* HER3-DXd becomes commercially available in the US and reimbursement is approved for the concerned indication of the Medical Access Program.
* Withdrawal of consent
* Pregnancy
* Physician discretion
* Death

ELIGIBILITY:
Inclusion Criteria - Initial Requests

* Signed informed consent.
* Male or female aged ≥18 years (or local regulatory requirements).
* Histologically or cytologically documented locally advanced or metastatic EGFRm NSCLC not amenable to curative surgery or radiation.
* Documentation of radiological disease progression whilst on/after receiving most recent treatment regimen for locally advanced or metastatic disease. Patients must have received both of the following:

  1. Prior treatment with any EGFR TKI, with at least one of them being osimertinib. Patients receiving an EGFR TKI at the time of signing informed consent should continue to take the EGFR TKI until 5 days prior to the first infusion of HER3 DXd.
  2. Systemic therapy with at least 1 PBC regimen.
* Documentation of an EGFR-activating mutation detected from tumor tissue or blood (exon 19 deletion or L858R mutation).
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at the time of entering the Medical Access Program.
* Adequate levels of bone marrow reserve and organ function, based on local laboratory data, within 14 days prior to the first HER3-DXd infusion as specified in the MAP protocol.
* Female patients of childbearing potential must have a negative urine or serum pregnancy test at the time of entering the Medical Access Program and must be willing to use highly effective contraception during the treatment period and for at least 7 months following the last dose of HER3-DXd. Additionally, female patients must agree to not donate, or retrieve for their own use, eggs from the time of entering the Medical Access Program and throughout the treatment period, and for at least 7 months after the final HER3-DXd administration. Male patients with female partners who are able to become pregnant must be willing to use a highly effective form of contraception or avoid intercourse during the treatment period and for at least 4 months following the last dose of HER3- DXd. Additionally, male patients must agree not freeze or donate sperm from time of entering the Medical Access Program and throughout the treatment period, and for at least 4 months after final dose of HER3- DXd.
* Life expectancy of >3 months as determined by the treating physician.

Inclusion Criteria - Resupply Requests

* Treating physician must confirm that the patient is deriving continued benefit from treatment.
* Treating physician must confirm that all required safety information has been reported as per local laws/regulations.

Exclusion Criteria - Initial Requests

* Patient is currently participating in or is in follow up for any Daiichi Sankyo ADC clinical trial including the HERTHENA-Lung02 'Trial of Patritumab Deruxtecan Initiated in Patients with EGFR-Mutated Metastatic Non-Small Cell Lung Cancer' (NCT05338970).
* Patient has previous or current histologic or cytologic evidence of small cell OR combined small cell/non-small cell disease in the archival tumor tissue or pre treatment tumor biopsy.
* Patient has any history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at the time of entering the Medical Access Program.
* Patient has clinically severe respiratory compromise (based on treating physician's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to: a) any underlying pulmonary disorder, b) any autoimmune, connective tissue or inflammatory disorders, OR c) prior complete pneumonectomy.
* Inadequate washout period prior to the first HER3-DXd infusion as specified in protocol.
* Clinically significant unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) Grade ≤1 or baseline. Patients with chronic Grade 2 toxicities may be eligible at the discretion of the treating physician after consultation with the designated Sponsor Medical Reviewer.
* Patient has clinically significant and/or uncontrolled cardiovascular disease prior to the first HER3-DXd infusion.
* Active hepatitis B virus (HBV) and/or hepatitis C virus infection, such as those with serologic evidence of viral infection within 28 days of the first HER3-DXd infusion.
* Human immunodeficiency virus (HIV) infection that is not well controlled as specified in the protocol.
* History of hypersensitivity to either the drug substance or any excipients in HER3-DXd.
* Female patient who is pregnant, breast-feeding, or intending to become pregnant.
* Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the treating physician's opinion, could affect the safety of the patient.
* Clinically significant corneal disease.
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection. Note: Patients with localized fungal infections of skin or nails are eligible.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Program Team Lead, Study Director — Daiichi Sankyo
Locations (21):
- United States (21):
  - Highlands Oncology, Springdale, Arkansas
  - Southern California Permanente Medical Group, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Advent Health, Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Block Medical Center, Skokie, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Karmanos Cancer Institute (Barbara Ann Karmanos Cancer Hospital), Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Washington University, St Louis, Missouri
  - Overlook Medical Center, Summit, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Kettering Health Cancer Center, New York, New York
  - The Mount Sinai Hospital- (Icahn School of Medicine), New York, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - The Kaiser Permanente Medical Group, Portland, Oregon
  - Texas Oncology, Pearland, Texas
  - Peace Health, Bellingham, Washington